CLINICAL TRIAL: NCT05976893
Title: Study on the Composite Endpoint Event of PCSK9 Inhibitor in Patients With Very High Risk of ASCVD and Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xiang Xie (Other)
Collaborators: Xinjiang Medical University (Other)
Responsible Party: Sponsor-Investigator, Xiang Xie, Principal Investigator, Xinjiang Medical University
Organization: Xinjiang Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PICVDAC
Record Dates: First submitted 2023-07-21; First posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-07

CONDITIONS: ASCVD; Atherosclerotic Cardiovascular Disease; Proprotein Convertase Subtilisin/Kexin Type 9 Inhibitor; Cancer
Keywords: ASCVD; cancer; PCSK9
MeSH Terms: conditions — Atherosclerosis; Neoplasms | interventions — evolocumab; Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Intervention Model Description: patients with very high risk of ASCVD and cancer
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- the PCSK9 inhibitor plus statin therapy (Experimental): Patients with very high risk of ASCVD and cancer are treated with moderate intensity statin daily and evolocumab (420 mg) every 4 weeks throughout the study period.
  Interventions: Drug: Evolocumab; Drug: Statin
- the statin alone therapy (Other): Patients with very high risk of ASCVD and cancer are treated with moderate intensity statin daily throughout the study period.
  Interventions: Drug: Statin

INTERVENTIONS:
Drug: Evolocumab — Evolocuma:420 mg every 4 weeks
  Other Names: Repatha
  Arms: the PCSK9 inhibitor plus statin therapy
Drug: Statin — The moderate intensity statins used during the study are one of atorvastatin 10-20mg qd, resuvastatin 5-10mg qd, and xuezhikang 0.6g bid (statin intolerance).

SUMMARY:
This study is a prospective, randomized, open-label, and single center trial. To evaluate the effect of treatment with PCSK9 inhibitor on the risk for cardiovascular death, recurrent unstable angina, myocardial infarction, stroke, or coronary revascularization in patients with very high risk of atherosclerotic cardiovascular disease (ASCVD) and cancer.

DETAILED DESCRIPTION:
Subjects will be randomly assigned in a 1:1 ratio to receive subcutaneous injections of PCSK9 inhibitor (evolocumab:420 mg every 4 weeks) plus moderate intensity statin therapy or the statin alone therapy. After randomization, patients will come to the hospital every 4 weeks to collect relevant laboratory results and clinical outcomes, and be detected by echocardiography and carotid ultrasound every 12 weeks until the end of follow-up at week 48 or the occurrence of an endpoint event. The entire study is expected to be conducted for 3 years, with a recruitment period of 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 to ≤ 80 years of age
* Patients with very high risk of ASCVD (with any of the following):

  1. Documented ASCVD, either clinical or unequivocal on imaging. Documented ASCVD includes previous acute coronary syndrome (ACS), stable angina, coronary revascularization (percutaneous coronary intervention, coronary artery bypass graft, and other arterial revascularization procedures), stroke and transient ischemic attack (TIA), and peripheral arterial disease. Unequivocally documented ASCVD on imaging includes those findings that are known to be predictive of clinical events, such as significant plaque on coronary angiography or computed tomography (CT) scan (multivessel coronary disease with two major epicardial arteries having >50% stenosis), or on carotid ultrasound.
  2. Diabetes mellitus (DM) with target organ damage, or at least three major risk factors, or early onset of type 1 diabetes mellitus (T1DM) of long duration (>20 years).
* Patients have been diagnosed with cancer through histopathology and have a life expectancy of more than 1 year
* Fasting low-density lipoprotein cholesterol (LDL-C) ≥ 1.8 mmol/L or non-high-density lipoprotein cholesterol (non HDL-C) > 2.6 mmol/L
* Participate voluntarily and sign an informed consent
* Negative serum Pregnancy test (in women with fertility potential)

Exclusion Criteria:

* Pregnant and lactating women
* During the study period and within 3 months of receiving the last dose of the study drug, women with fertility intentions and men unwilling to use effective contraceptive methods
* New York Heart Association (NYHA) class III or IV, or last known left ventricular ejection fraction < 30%
* Uncontrolled hypertension, defined as systolic blood pressure ≥ 180 mmHg and/or diastolic blood pressure ≥ 110 mmHg
* Plan for coronary revascularization or other cardiac surgery in recent (within 3 months after randomization)
* Severe renal insufficiency, defined as estimated glomerular filtration rate (eGRF) < 30ml/min/1.73m2 or Serum creatinine (Scr) > 221 umol/L
* Severe liver dysfunction, defined as an increase in alanine aminotransferase (ALT) or aspartate aminotransferase (AST) more than 3 times above the upper limit of normal
* Have used PCSK9 inhibitors within 3 months before enrollment, or have a history of severe allergic reactions to PCSK9 inhibitors
* Severe infections requiring intravenous antibiotics
* HIV-positive or history of acquired immunodeficiency syndrome (AIDS)
* With cognitive impairment or psychiatric illnesses
* Participating in other trials

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 620 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Major cardiovascular adverse events | From date of randomization until the date of first documented endpoint or date of completion of follow-up, whichever came first, assessed up to 48 weeks
  Major cardiovascular adverse events include cardiovascular death, recurrent unstable angina, myocardial infarction, stroke, and coronary revascularization

SECONDARY OUTCOMES:
All cause death | From date of randomization until the date of first documented endpoint or date of completion of follow-up, whichever came first, assessed up to 48 weeks
  All cause death
Composite end points | From date of randomization until the date of first documented endpoint or date of completion of follow-up, whichever came first, assessed up to 48 weeks
  Composite end points include cardiogenic shock, cardiac arrest, malignant arrhythmia, heart failure, Non-coronary revascularization
The compliance rate of lipid control | From date of randomization until the date of first documented endpoint or date of completion of follow-up, whichever came first, assessed up to 48 weeks
  Main indicator: LDL-C decreased to below 1.4 mmol/L and decreased by more than 50% from baseline; secondary indicator: non HDL-C<2.2 mmol/L;
The changes of carotid plaque | From date of randomization until the date of first documented endpoint or date of completion of follow-up, whichever came first, assessed up to 48 weeks
  By carotid ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Xie, PhD, Principal Investigator — First Affiliated Hospital of Xinjiang Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhou M, Wang H, Zeng X, Yin P, Zhu J, Chen W, Li X, Wang L, Wang L, Liu Y, Liu J, Zhang M, Qi J, Yu S, Afshin A, Gakidou E, Glenn S, Krish VS, Miller-Petrie MK, Mountjoy-Venning WC, Mullany EC, Redford SB, Liu H, Naghavi M, Hay SI, Wang L, Murray CJL, Liang X. Mortality, morbidity, and risk factors in China and its provinces, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2019 Sep 28;394(10204):1145-1158. doi: 10.1016/S0140-6736(19)30427-1. Epub 2019 Jun 24. PMID 31248666
- [Result] Xia C, Dong X, Li H, Cao M, Sun D, He S, Yang F, Yan X, Zhang S, Li N, Chen W. Cancer statistics in China and United States, 2022: profiles, trends, and determinants. Chin Med J (Engl). 2022 Feb 9;135(5):584-590. doi: 10.1097/CM9.0000000000002108. PMID 35143424
- [Result] Zeng H, Chen W, Zheng R, Zhang S, Ji JS, Zou X, Xia C, Sun K, Yang Z, Li H, Wang N, Han R, Liu S, Li H, Mu H, He Y, Xu Y, Fu Z, Zhou Y, Jiang J, Yang Y, Chen J, Wei K, Fan D, Wang J, Fu F, Zhao D, Song G, Chen J, Jiang C, Zhou X, Gu X, Jin F, Li Q, Li Y, Wu T, Yan C, Dong J, Hua Z, Baade P, Bray F, Jemal A, Yu XQ, He J. Changing cancer survival in China during 2003-15: a pooled analysis of 17 population-based cancer registries. Lancet Glob Health. 2018 May;6(5):e555-e567. doi: 10.1016/S2214-109X(18)30127-X. PMID 29653628
- [Result] Miller KD, Nogueira L, Devasia T, Mariotto AB, Yabroff KR, Jemal A, Kramer J, Siegel RL. Cancer treatment and survivorship statistics, 2022. CA Cancer J Clin. 2022 Sep;72(5):409-436. doi: 10.3322/caac.21731. Epub 2022 Jun 23. PMID 35736631
- [Result] Lyon AR, Lopez-Fernandez T, Couch LS, Asteggiano R, Aznar MC, Bergler-Klein J, Boriani G, Cardinale D, Cordoba R, Cosyns B, Cutter DJ, de Azambuja E, de Boer RA, Dent SF, Farmakis D, Gevaert SA, Gorog DA, Herrmann J, Lenihan D, Moslehi J, Moura B, Salinger SS, Stephens R, Suter TM, Szmit S, Tamargo J, Thavendiranathan P, Tocchetti CG, van der Meer P, van der Pal HJH; ESC Scientific Document Group. 2022 ESC Guidelines on cardio-oncology developed in collaboration with the European Hematology Association (EHA), the European Society for Therapeutic Radiology and Oncology (ESTRO) and the International Cardio-Oncology Society (IC-OS). Eur Heart J. 2022 Nov 1;43(41):4229-4361. doi: 10.1093/eurheartj/ehac244. No abstract available. PMID 36017568
- [Result] Bergom C, Bradley JA, Ng AK, Samson P, Robinson C, Lopez-Mattei J, Mitchell JD. Past, Present, and Future of Radiation-Induced Cardiotoxicity: Refinements in Targeting, Surveillance, and Risk Stratification. JACC CardioOncol. 2021 Sep 21;3(3):343-359. doi: 10.1016/j.jaccao.2021.06.007. eCollection 2021 Sep. PMID 34604796
- [Result] Bharadwaj A, Potts J, Mohamed MO, Parwani P, Swamy P, Lopez-Mattei JC, Rashid M, Kwok CS, Fischman DL, Vassiliou VS, Freeman P, Michos ED, Mamas MA. Acute myocardial infarction treatments and outcomes in 6.5 million patients with a current or historical diagnosis of cancer in the USA. Eur Heart J. 2020 Jun 14;41(23):2183-2193. doi: 10.1093/eurheartj/ehz851. PMID 31800032
- [Result] Gevaert SA, Halvorsen S, Sinnaeve PR, Sambola A, Gulati G, Lancellotti P, Van Der Meer P, Lyon AR, Farmakis D, Lee G, Boriani G, Wechalekar A, Okines A, Asteggiano R. Evaluation and management of cancer patients presenting with acute cardiovascular disease: a Consensus Document of the Acute CardioVascular Care (ACVC) association and the ESC council of Cardio-Oncology-Part 1: acute coronary syndromes and acute pericardial diseases. Eur Heart J Acute Cardiovasc Care. 2021 Oct 27;10(8):947-959. doi: 10.1093/ehjacc/zuab056. PMID 34453829
- [Result] Mach F, Baigent C, Catapano AL, Koskinas KC, Casula M, Badimon L, Chapman MJ, De Backer GG, Delgado V, Ference BA, Graham IM, Halliday A, Landmesser U, Mihaylova B, Pedersen TR, Riccardi G, Richter DJ, Sabatine MS, Taskinen MR, Tokgozoglu L, Wiklund O; ESC Scientific Document Group. 2019 ESC/EAS Guidelines for the management of dyslipidaemias: lipid modification to reduce cardiovascular risk. Eur Heart J. 2020 Jan 1;41(1):111-188. doi: 10.1093/eurheartj/ehz455. No abstract available. PMID 31504418
- [Result] Sabatine MS, Giugliano RP, Keech AC, Honarpour N, Wiviott SD, Murphy SA, Kuder JF, Wang H, Liu T, Wasserman SM, Sever PS, Pedersen TR; FOURIER Steering Committee and Investigators. Evolocumab and Clinical Outcomes in Patients with Cardiovascular Disease. N Engl J Med. 2017 May 4;376(18):1713-1722. doi: 10.1056/NEJMoa1615664. Epub 2017 Mar 17. PMID 28304224
- [Result] Sabatine MS, Giugliano RP, Wiviott SD, Raal FJ, Blom DJ, Robinson J, Ballantyne CM, Somaratne R, Legg J, Wasserman SM, Scott R, Koren MJ, Stein EA; Open-Label Study of Long-Term Evaluation against LDL Cholesterol (OSLER) Investigators. Efficacy and safety of evolocumab in reducing lipids and cardiovascular events. N Engl J Med. 2015 Apr 16;372(16):1500-9. doi: 10.1056/NEJMoa1500858. Epub 2015 Mar 15. PMID 25773607
- [Result] Schwartz GG, Steg PG, Szarek M, Bhatt DL, Bittner VA, Diaz R, Edelberg JM, Goodman SG, Hanotin C, Harrington RA, Jukema JW, Lecorps G, Mahaffey KW, Moryusef A, Pordy R, Quintero K, Roe MT, Sasiela WJ, Tamby JF, Tricoci P, White HD, Zeiher AM; ODYSSEY OUTCOMES Committees and Investigators. Alirocumab and Cardiovascular Outcomes after Acute Coronary Syndrome. N Engl J Med. 2018 Nov 29;379(22):2097-2107. doi: 10.1056/NEJMoa1801174. Epub 2018 Nov 7. PMID 30403574
- [Result] Cannon CP, Blazing MA, Giugliano RP, McCagg A, White JA, Theroux P, Darius H, Lewis BS, Ophuis TO, Jukema JW, De Ferrari GM, Ruzyllo W, De Lucca P, Im K, Bohula EA, Reist C, Wiviott SD, Tershakovec AM, Musliner TA, Braunwald E, Califf RM; IMPROVE-IT Investigators. Ezetimibe Added to Statin Therapy after Acute Coronary Syndromes. N Engl J Med. 2015 Jun 18;372(25):2387-97. doi: 10.1056/NEJMoa1410489. Epub 2015 Jun 3. PMID 26039521
- [Result] Hu J, La Vecchia C, de Groh M, Negri E, Morrison H, Mery L; Canadian Cancer Registries Epidemiology Research Group. Dietary cholesterol intake and cancer. Ann Oncol. 2012 Feb;23(2):491-500. doi: 10.1093/annonc/mdr155. Epub 2011 May 4. PMID 21543628
- [Result] Hao Q, Aertgeerts B, Guyatt G, Bekkering GE, Vandvik PO, Khan SU, Rodondi N, Jackson R, Reny JL, Al Ansary L, Van Driel M, Assendelft WJJ, Agoritsas T, Spencer F, Siemieniuk RAC, Lytvyn L, Heen AF, Zhao Q, Riaz IB, Ramaekers D, Okwen PM, Zhu Y, Dawson A, Ovidiu MC, Vanbrabant W, Li S, Delvaux N. PCSK9 inhibitors and ezetimibe for the reduction of cardiovascular events: a clinical practice guideline with risk-stratified recommendations. BMJ. 2022 May 4;377:e069066. doi: 10.1136/bmj-2021-069066. PMID 35508320
- [Result] Gong Y, Li X, Ma X, Yu H, Li Y, Chen J, Zhang G, Wang B, Qi X, Meng H, Wang X, Mu J, Hu X, Wang J, Liu S, Liu G, Yang Z, Zhou Y, Kong X, Yan Y, Wang C, Wang JA, Wang L, Fu G, Wei L, Peng D, Zhang S, Li R, Mao A, Bian R, Tang W, Ran Y, Jiang J, Huo Y. Lipid goal attainment in post-acute coronary syndrome patients in China: Results from the 6-month real-world dyslipidemia international study II. Clin Cardiol. 2021 Nov;44(11):1575-1585. doi: 10.1002/clc.23725. Epub 2021 Oct 15. PMID 34651329
- [Result] Schludi B, Giugliano RP, Sabatine MS, Raal FJ, Teramoto T, Koren MJ, Stein EA, Wang H, Monsalvo ML. Time-averaged low-density lipoprotein cholesterol lowering with evolocumab: Pooled analysis of phase 2 trials. J Clin Lipidol. 2022 Jul-Aug;16(4):538-543. doi: 10.1016/j.jacl.2022.05.069. Epub 2022 Jun 6. PMID 35760720
- [Result] Desai NR, Giugliano RP, Zhou J, Kohli P, Somaratne R, Hoffman E, Liu T, Scott R, Wasserman SM, Sabatine MS. AMG 145, a monoclonal antibody against PCSK9, facilitates achievement of national cholesterol education program-adult treatment panel III low-density lipoprotein cholesterol goals among high-risk patients: an analysis from the LAPLACE-TIMI 57 trial (LDL-C assessment with PCSK9 monoclonal antibody inhibition combined with statin thErapy-thrombolysis in myocardial infarction 57). J Am Coll Cardiol. 2014 Feb 11;63(5):430-3. doi: 10.1016/j.jacc.2013.09.048. Epub 2013 Oct 23. PMID 24161333
- [Result] O'Donoghue ML, Giugliano RP, Wiviott SD, Atar D, Keech A, Kuder JF, Im K, Murphy SA, Flores-Arredondo JH, Lopez JAG, Elliott-Davey M, Wang B, Monsalvo ML, Abbasi S, Sabatine MS. Long-Term Evolocumab in Patients With Established Atherosclerotic Cardiovascular Disease. Circulation. 2022 Oct 11;146(15):1109-1119. doi: 10.1161/CIRCULATIONAHA.122.061620. Epub 2022 Aug 29. PMID 36031810
- [Result] American Diabetes Association Professional Practice Committee. 10. Cardiovascular Disease and Risk Management: Standards of Medical Care in Diabetes-2022. Diabetes Care. 2022 Jan 1;45(Suppl 1):S144-S174. doi: 10.2337/dc22-S010. PMID 34964815
- [Result] China Cholesterol Education Program (CCEP) Working Committee; Atherosclerosis Thrombosis Prevention and Control Subcommittee of Chinese International Exchange and Promotion Association for Medical and Healthcare; Cardiovascular Disease Subcommittee of China Association of Gerontology and Geriatrics; Atherosclerosis Professional Committee of Chinese College of Cardiovascular Physicians. [China cholesterol education program (CCEP) expert advice for the management of dyslipidaemias to reduce cardiovascular risk (2019)]. Zhonghua Nei Ke Za Zhi. 2020 Jan 1;59(1):18-22. doi: 10.3760/cma.j.issn.0578-1426.2020.01.003. Chinese. PMID 31887831
- [Result] Atherosclerosis and Coronary Heart Disease Working Group of Chinese Society of Cardiology; Editorial Board of Chinese Journal of Cardiology. [Chinese expert consensus on lipid management of very high-risk atherosclerotic cardiovascular disease patients]. Zhonghua Xin Xue Guan Bing Za Zhi. 2020 Apr 24;48(4):280-286. doi: 10.3760/cma.j.cn112148-20200121-00036. Chinese. PMID 32370478
- [Result] Integrative Cardio-Oncology Society of China Anti-Cancer Association. [Chinese expert consensus on lipid management in patients with malignancy]. Zhonghua Zhong Liu Za Zhi. 2021 Oct 23;43(10):1043-1053. doi: 10.3760/cma.j.cn112152-20210415-00321. Chinese. PMID 34695894
- [Result] In China TWCOTROCHAD, Hu SS. Report on cardiovascular health and diseases in China 2021: an updated summary. J Geriatr Cardiol. 2023 Jun 28;20(6):399-430. doi: 10.26599/1671-5411.2023.06.001. PMID 37416519